CLINICAL TRIAL: NCT04593797
Title: The Accuracy of Ultrasound Derived Carotid, Femoral and Brachial Artery Compared to Conventional Intra-vascular Methods Flow-related Parameters
Brief Title: Echo FLOW Versus (Non-)Invasive Haemodynamics
Acronym: EFLOW
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, A.P.J. Vlaar, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL64436.018.17
Record Dates: First submitted 2020-09-29; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Cardiac Output, Low; Cardiac Output, High
MeSH Terms: conditions — Cardiac Output, Low; Cardiac Output, High | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing major upper abdominal surgery: major open upper abdominal surgery eg pancreatic, liver surgery
  Interventions: Diagnostic Test: carotid blood flow measurement with ultrasound

INTERVENTIONS:
Diagnostic Test: carotid blood flow measurement with ultrasound — carotid blood flow measurement with ultrasound vs transpulmonary thermodilution calibrated continuous cardiac output measurements
  Other Names: transpulmonary thermodilution calibrated continuous cardiac output measurements

SUMMARY:
Rationale: Diligent fluid management is instrumental to improve postoperative outcome, cost and quality of care.

Objective: To determine the accuracy of brachial, femoral and carotid blood flow measurement with ultrasound compared to intermittent transpulmonary thermodilution cardiac output measurement, invasive and non-invasive pulse-contour analysis.

Study design: Observational study - Prospective clinical non-intervention measurement study.

Study population: Adult ASA 1-2 patients, scheduled for open upper GI surgery Intervention (if applicable): Not applicable. We will perform non-invasive ultrasound measurements of the femoral, carotid and brachial blood flow right before induction and under anaesthesia.

Main study parameters/endpoints: Femoral, carotid and brachial blood flow determined by ultrasound and blood flow variation and the accuracy compared to transpulmonary thermodilution cardiac output, stroke volume variation, and pulse-contour analysis derived cardiac output (invasive or non-invasive) at the following time points during surgery; (limited for femoral site as it cannot be measured during surgery): (1) before induction of anaesthesia, (2) after induction, (3) 15 minutes after start of surgery, (4) before and (5) after (1-2 minutes) a fluid bolus, (6) before and (7) after start of vasopressors, (8) before and (9) after Trendelenburg position and (10) after surgery before end of anaesthesia (figure 1). A fluid bolus will be performed as part of standard care (goal-directed fluid therapy). The vasopressor and Trendelenburg position time points are optional measurements. We will also measure (continuous) invasive femoral blood pressure (SBP, DBP, MAP), non-invasive blood pressure, SVV, central venous pressure (when available), heart rate, SpO2, PFI, etCO2.

ELIGIBILITY:
Inclusion Criteria:

* Elective open GI surgery
* Invasive arterial blood pressure monitoring
* Informed consent

Exclusion Criteria:

* Significant stenosis > 30% or abnormal anatomy of aortic, femoral, carotid or brachial artery
* Cerebrovascular accident
* Atrial fibrillation
* COPD stage 3-4
* Lobectomy / pneumectomy
* Active pneumonia
* Cardiac failure
* Severe heart valve regurgitation or stenosis
* Not able to measure brachial or carotid artery blood flow during surgery
* Contra-indications for femoral arterial catheter placement (e.g., vascular graft)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, scheduled for open upper GI surgery with a American Society of Anaesthesiologist score of 1 to 2
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Cardiac output | baseline
  blood flow determined by ultrasound and the accuracy compared to transpulmonary thermodilution calibrated continuous cardiac output

SECONDARY OUTCOMES:
Cardiac output change | change from baseline cardiac output 1 minute after intervention (fluid challenge, vasopressor administration, or Trendelenburg)
  Change in blood flow compared to change in cardiac output

CONTACTS AND LOCATIONS:
Overall Officials: A.P. Vlaar, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Academisch Medisch Centrum - Universiteit van Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Plan to make individual available upon request